CLINICAL TRIAL: NCT01038934
Title: Evaluation of Genomic DNA of Oral Cytobrush in Three Means Conservation
Brief Title: DNA of Oral Cytobrush in Three Means Conservation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Glauco Issamu Miyahara/ Professor, School of Dentistry, Sao Paulo State University, Unesp, Araçatuba/SP
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: upeclin/FOA-Unesp-04
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-12

CONDITIONS: Healthy
Keywords: Buccal Mucosa; DNA; Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- buccal cytobrhsh (Experimental): healthy young
  Interventions: Procedure: samples collected by buccal cytobrush

INTERVENTIONS:
Procedure: samples collected by buccal cytobrush

SUMMARY:
The aim of this study is to analyze genomic DNA of buccal cytobrush stored in three means conservation.

DETAILED DESCRIPTION:
Blood samples are an excellent source of large amounts of genomic DNA. However, alternative sources are often needed in epidemiological studies because of difficulties in obtaining blood samples.

ELIGIBILITY:
Inclusion Criteria:

* healthy young

Exclusion Criteria:

* none

Ages: 20 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2006-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glauco I Miyahara, Professor, Principal Investigator — Univ. Estadual Paulista
Locations (1):
- School of Dentistry, Sao Paulo State University, Unesp, Araçatuba/SP, Araçatuba, São Paulo, Brazil